CLINICAL TRIAL: NCT04539262
Title: A Phase 1b/2a Study in Participants With Early Stage COVID-19 to Evaluate the Safety, Efficacy, and Pharmacokinetics of Remdesivir Administered by Inhalation
Brief Title: Study in Participants With Early Stage Coronavirus Disease 2019 (COVID-19) to Evaluate the Safety, Efficacy, and Pharmacokinetics of Remdesivir Administered by Inhalation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-553-9020
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Remdesivir (RDV), Part A (Experimental): Participants will receive inhaled RDV 31 mg administered daily for 5 days.
  Interventions: Drug: Remdesivir (RDV)
- RDV + Placebo, Part A (Experimental): Participants will receive inhaled RDV 31 mg administered daily for 3 days followed by placebo to match RDV daily for 2 days.
  Interventions: Drug: Remdesivir (RDV); Drug: Placebo
- Placebo, Part A (Placebo Comparator): Participants will receive placebo to match inhaled RDV in Part A daily for 5 days.
  Interventions: Drug: Placebo
- RDV, Part B (Experimental): Participants will receive inhaled RDV 62 mg administered daily for up to 5 days.
  Interventions: Drug: Remdesivir (RDV)
- RDV + Placebo, Part B (Experimental): Participants will receive inhaled RDV 62 mg administered daily for up to 3 days followed by placebo to match RDV daily for 2 days.
  Interventions: Drug: Remdesivir (RDV); Drug: Placebo
- Placebo, Part B (Placebo Comparator): Participants will receive placebo to match inhaled RDV in Part B daily for 5 days.
  Interventions: Drug: Placebo
- RDV, Part C (Experimental): Participants will receive inhaled RDV 39 mg administered daily for 5 days.
  Interventions: Drug: Remdesivir (RDV)
- Placebo, Part C (Placebo Comparator): Participants will receive placebo to match inhaled RDV in Part C daily for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remdesivir (RDV) — Administered as an aerosolized solution
  Other Names: GS-5734™
  Arms: RDV + Placebo, Part A; RDV + Placebo, Part B; RDV, Part B; RDV, Part C; Remdesivir (RDV), Part A
Drug: Placebo — Administered as an aerosolized solution
  Arms: Placebo, Part A; Placebo, Part B; Placebo, Part C; RDV + Placebo, Part A; RDV + Placebo, Part B

SUMMARY:
The primary objective of this study is to characterize the impact of inhaled remdesivir (RDV) on severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) viral load in participants with early stage coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
This study will have multiple parts: Part A, Part B, and Part C. Part B will be conducted if supported by evaluation in healthy volunteers in another Phase 1a Gilead study (GS-US-553-9018). Participants in Part C will be enrolled after review of preliminary safety and available efficacy data from Parts A and B through at least Day 7.

GS-US-553-9018 is a Phase 1a randomized, blinded, placebo-controlled, single- and multiple-dose study in healthy volunteers to evaluate the safety, tolerability, and pharmacokinetics of remdesivir administered by inhalation.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent
* SARS-CoV-2 infection first confirmed by polymerase chain reaction (PCR) (Parts A and B) or by nucleic acid testing or direct antigen testing (Part C) with sample collected ≤ 4 days prior to randomization
* COVID-19 symptom onset ≤ 7 days prior to randomization
* Oxygen saturation as measured by pulse oximetry (SpO2) > 94% on room air

Key Exclusion Criteria:

* Ongoing or prior participation in any other clinical trial of an experimental vaccine or treatment for COVID-19
* Prior or current hospitalization for COVID-19 or need for hospitalization
* Treatment of COVID-19 with other agents with actual or possible direct antiviral activity against SARS-CoV-2 including intravenous (IV) RDV or administration of any SARS-CoV-2 (or COVID-19) vaccine

  * Participants chronically administered chloroquine or hydroxychloroquine for any reason are to be excluded
* Requiring oxygen supplementation
* Positive pregnancy test
* Breastfeeding female
* Known hypersensitivity to the study treatment, its metabolites, or formulation excipient
* Pre-existing pulmonary conditions such as chronic obstructive pulmonary disease or asthma (Parts A and B only)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (28):
- United States (28):
  - The Institute for Liver Health, Mesa, Arizona
  - The Institute for Liver Health, Tucson, Arizona
  - Franco Felizarta, MD, Bakersfield, California
  - Aurora FDRC Inc., Costa Mesa, California
  - Elevated Health, Huntington Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Western Clinical Research, Placentia, California
  - UC Davis Health/Medical Center, Sacramento, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Research in Miami, Inc., Hialeah, Florida
  - Evolution Clinical Trials, Inc., Hialeah Gardens, Florida
  - Optimus U Corporation, Miami, Florida
  - L & C Professional Medical Research Institute, Miami, Florida
  - Westchester Research Center at Westchester General Hospital, Miami, Florida
  - MedBio Trials, Miami, Florida
  - Nuovida Research Center, Corp, Miami, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Triple O Research Institute, PA, West Palm Beach, Florida
  - Family Care Research, Boise, Idaho
  - CTU Covid Research Center, New Orleans, Louisiana
  - STAT Research, Vandalia, Ohio
  - Inquest Clinical Research, Baytown, Texas
  - DFW Clinical Research, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - PCP for Life-Tidwell, Houston, Texas
  - Providence Regional Medical Center Everett, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 14 September 2020. The last study visit occurred on 22 March 2021.
Pre-assignment Details: 168 participants were screened.
Groups:
- Remdesivir (RDV), Part A: Participants received inhaled remdesivir (RDV) 31 mg administered daily as an aerosolized solution by inhalation through facemask for 5 days.
- RDV + Placebo, Part A: Participants received inhaled RDV 31 mg administered daily as an aerosolized solution by inhalation through facemask for 3 days followed by placebo to match RDV daily for 2 days.
- Placebo, Part A: Participants received placebo to match inhaled RDV in Part A daily for 5 days.
- RDV, Part B: Participants received inhaled RDV 62 mg administered daily as an aerosolized solution by inhalation through facemask for 5 days.
- RDV + Placebo, Part B: Participants received inhaled RDV 62 mg administered daily as an aerosolized solution by inhalation through facemask for 3 days followed by placebo to match RDV daily for 2 days.
- Placebo, Part B: Participants received placebo to match inhaled RDV in Part B daily for 5 days.
- RDV, Part C: Participants received inhaled RDV 39 mg administered daily as an aerosolized solution by inhalation through mouth piece for 5 days.
- Placebo, Part C: Participants received placebo to match inhaled RDV in Part C daily for 5 days.
Period: Overall Study
Arm/Group | Remdesivir (RDV), Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Started | 12 | 13 | 12 | 12 | 12 | 13 | 62 | 20
Completed | 12 | 12 | 11 | 11 | 12 | 13 | 61 | 20
Not Completed | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized, Not treated | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study treatment.
Groups:
- RDV, Part A: Participants received inhaled RDV 31 mg administered daily as an aerosolized solution by inhalation through facemask for 5 days.
- Total: Total of all reporting groups
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20 | 154
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 10 | 11 | 9 | 12 | 10 | 12 | 55 | 15 | 134
  ≥ 60 years | 2 | 1 | 3 | 0 | 2 | 1 | 6 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 4 | 7 | 5 | 6 | 34 | 8 | 77
  Male | 4 | 7 | 8 | 5 | 7 | 7 | 27 | 12 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 3 | 2 | 6 | 4 | 40 | 14 | 78
  Not Hispanic or Latino | 6 | 9 | 9 | 10 | 4 | 9 | 21 | 6 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: Asian | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Race: Black | 0 | 0 | 0 | 0 | 1 | 1 | 12 | 2 | 16
    Race: White | 11 | 9 | 10 | 11 | 10 | 12 | 47 | 16 | 126
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Race: Not Permitted | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 5
    Race: Other | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
SARS-CoV-2 Viral load - Nasopharyngeal [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  log10 copies/mL
    number analyzed (Participants) | 12 | 11 | 12 | 10 | 10 | 13 | 57 | 18 | 143
    (all) | 7.29 (1.901) | 6.56 (1.065) | 6.81 (1.065) | 5.23 (1.980) | 6.41 (1.883) | 7.09 (1.288) | 5.69 (2.004) | 5.76 (1.839) | 6.14 (1.859)
SARS-CoV-2 Viral load - Oropharyngeal [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  log10 copies/mL
    number analyzed (Participants) | 11 | 11 | 12 | 11 | 10 | 12 | 57 | 18 | 142
    (all) | 5.69 (0.959) | 4.74 (1.225) | 5.57 (1.275) | 4.40 (1.772) | 5.16 (1.356) | 4.79 (1.377) | 4.38 (1.610) | 3.94 (1.203) | 4.64 (1.505)
SARS-CoV-2 Viral load - Saliva [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  log10 copies/mL
    number analyzed (Participants) | 10 | 11 | 9 | 11 | 10 | 13 | 59 | 19 | 142
    (all) | 5.56 (1.682) | 5.19 (1.312) | 4.77 (1.218) | 5.15 (2.048) | 4.77 (1.281) | 5.60 (1.074) | 4.93 (1.785) | 4.57 (1.559) | 5.00 (1.613)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average Change From Baseline in Nasopharyngeal Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load Through Day 7
Description: Time-weighted average change in SARS-CoV-2 viral load was defined as area under the concentration versus time curve (AUC) of viral load change divided by time between baseline through Day 7.
Time Frame: Baseline, Day 7
Population: Participants in the Nasopharyngeal Modified Full Analysis Set (mFAS) (all participants who were randomized into the study, had received at least 1 dose of study treatment and had positive SARS-CoV-2 viral load using nasopharyngeal swab sample at baseline [the result of 'No SARS-CoV-2 detected' was considered as negative]) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 11 | 11 | 8 | 10 | 13 | 44 | 16
log10 copies/mL | -2.04 (0.999) | -1.51 (0.812) | -1.24 (0.961) | -1.21 (1.108) | -1.42 (0.975) | -1.40 (0.796) | -1.91 (1.186) | -1.93 (1.284)
Statistical Analysis 1: Comparison: RDV, Part A vs Placebo, Part A; Test type: Superiority; p = 0.1117, ANCOVA — Least square (LS) Mean, Standard Error (SE), 95% CI and p-value were from Analysis of covariance (ANCOVA) with baseline viral load as a covariate; Least Square Mean Difference by Day 7 = -0.66, 95% CI 2-sided [-1.49 to 0.16], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: RDV + Placebo, Part A vs Placebo, Part A; Test type: Superiority; p = 0.3793, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.35, 95% CI 2-sided [-1.16 to 0.46], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: RDV, Part B vs Placebo, Part B; Test type: Superiority; p = 0.5248, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.24, 95% CI 2-sided [-1.00 to 0.52], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: RDV + Placebo, Part B vs Placebo, Part B; Test type: Superiority; p = 0.4610, ANCOVA; LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.25, 95% CI 2-sided [-0.94 to 0.44], Standard Error of Mean 0.34
Statistical Analysis 5: Comparison: RDV, Part C vs Placebo, Part C; Test type: Superiority; p = 0.5006, ANCOVA — LS Mean (SE), 95% CI and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.20, 95% CI 2-sided [-0.40 to 0.81], Standard Error of Mean 0.30

2. Primary Outcome: Time-weighted Average Change From Baseline in Oropharyngeal SARS-CoV-2 Viral Load Through Day 7
Description: Time-weighted average change in SARS-CoV-2 viral load was defined as AUC of viral load change divided by time between baseline through Day 7.
Time Frame: Baseline, Day 7
Population: Participants in the Oropharyngeal mFAS (all participants who were randomized into the study, had received at least 1 dose of study treatment and had positive SARS-CoV-2 viral load using oropharyngeal swab sample at baseline [the result of 'No SARS-CoV-2 detected' was considered as negative]) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 11 | 41 | 12
log10 copies/mL | -1.10 (0.856) | -0.55 (0.868) | -1.39 (1.036) | -1.14 (1.133) | -0.85 (1.164) | -0.70 (0.902) | -0.83 (1.073) | -0.46 (1.152)
Statistical Analysis 1: Comparison: RDV, Part A vs Placebo, Part A; Test type: Superiority; p = 0.3417, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.33, 95% CI 2-sided [-0.37 to 1.02], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: RDV + Placebo, Part A vs Placebo, Part A; Test type: Superiority; p = 0.1803, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.49, 95% CI 2-sided [-0.24 to 1.21], Standard Error of Mean 0.35
Statistical Analysis 3: Comparison: RDV, Part B vs Placebo, Part B; Test type: Superiority; p = 0.1233, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.55, 95% CI 2-sided [-1.27 to 0.16], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: RDV + Placebo, Part B vs Placebo, Part B; Test type: Superiority; p = 0.8203, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.08, 95% CI 2-sided [-0.64 to 0.80], Standard Error of Mean 0.35
Statistical Analysis 5: Comparison: RDV, Part C vs Placebo, Part C; Test type: Superiority; p = 0.6458, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.12, 95% CI 2-sided [-0.65 to 0.41], Standard Error of Mean 0.26

3. Primary Outcome: Time-weighted Average Change From Baseline in Saliva SARS-CoV-2 Viral Load Through Day 7
Description: as for outcome 2
Time Frame: Baseline, Day 7
Population: Participants in the saliva mFAS (all participants who were randomized into the study, had received at least 1 dose of study treatment and had positive SARS-CoV-2 viral load using saliva swab sample at baseline [the result of 'No SARS-CoV-2 detected' was considered as negative]) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 9 | 12 | 44 | 16
log10 copies/mL | -0.80 (0.469) | -1.27 (0.877) | -0.49 (1.148) | -1.09 (1.497) | -0.61 (0.676) | -0.93 (0.678) | -1.25 (0.977) | -1.01 (1.096)
Statistical Analysis 1: Comparison: RDV, Part A vs Placebo, Part A; Test type: Superiority; p = 0.5951, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.22, 95% CI 2-sided [-1.05 to 0.61], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: RDV + Placebo, Part A vs Placebo, Part A; Test type: Superiority — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; p = 0.0872, ANCOVA; LS Mean Difference by Day 7 = -0.71, 95% CI 2-sided [-1.54 to 0.11], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: RDV, Part B vs Placebo, Part B; Test type: Superiority; p = 0.6031, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = -0.19, 95% CI 2-sided [-0.94 to 0.56], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: RDV + Placebo, Part B vs Placebo, Part B; Test type: Superiority; p = 0.7578, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.12, 95% CI 2-sided [-0.64 to 0.87], Standard Error of Mean 0.37
Statistical Analysis 5: Comparison: RDV, Part C vs Placebo, Part C; Test type: Superiority; p = 0.8846, ANCOVA — LS Mean (SE), 95% CI, and p-value were from ANCOVA with baseline viral load as a covariate; LS Mean Difference by Day 7 = 0.04, 95% CI 2-sided [-0.48 to 0.56], Standard Error of Mean 0.26

4. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a study drug, which did not necessarily have a causal relationship with the treatment. AE was therefore any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug. TEAEs: AE with an onset date on or after the study drug start date and no later than 30 days after study drug stop date; or any AE leading to study drug discontinuation.
Time Frame: First dose date up to 5 days plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20
percentage of participants | 58.3 | 58.3 | 41.7 | 33.3 | 58.3 | 38.5 | 42.6 | 25.0

5. Secondary Outcome: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities as Per Severity Grade
Description: Treatment-emergent laboratory abnormalities were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 July 2017. Laboratory abnormalities were graded as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening). Percentage of participants with any severity grade were reported.
Time Frame: First dose date up to 5 days plus 30 days
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 11 | 11 | 12 | 13 | 61 | 20
percentage of participants | 58.3 | 91.7 | 63.6 | 63.6 | 83.3 | 61.5 | 68.9 | 75.0

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events Leading to Study Treatment Discontinuation
Time Frame: First dose date up to 5 days plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20
percentage of participants | 0 | 0 | 8.3 | 0 | 0 | 0 | 1.6 | 0

7. Secondary Outcome: Number of Participants With All-Cause Medically Attended Visits (MAVs) or Death by Day 28
Description: The composite outcome of all-cause MAVs (medical visits attended in person by the participant and a health care professional) or all-cause death by Study Day 28 were estimated using Kaplan-Meier methods by treatment group.
Time Frame: Randomization up to Day 28
Population: Participants in the Full Analysis Set (all participants who were randomized into the study, and had received at least 1 dose of study treatment) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20
Participants | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With COVID-19 Related MAVs or Death by Day 28
Description: The composite outcome of COVID-19 related MAVs (medical visits attended in person by the participant and a health care professional) or all-cause death by Study Day 28 were estimated using Kaplan-Meier methods by treatment group.
Time Frame: Randomization up to Day 28
Population: Participants in the Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20
Participants | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Hospitalization by Day 28
Description: The composite of all-cause hospitalization was estimated using Kaplan-Meier methods by treatment group.
Time Frame: Day 1 up to Day 28
Population: Participants in the Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 13 | 61 | 20
Participants | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0

10. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUC0-24h of Remdesivir (RDV) and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: AUC0-24h was defined as the concentration of drug over time between time 0 to time 24 hours. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: Sparse PK: Day 1 (end of nebulization) and Day 3 (predose and end of nebulization); Intensive PK: Day 1 and Day 3 or Day 5 (0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization); Nebulization duration: 17-34 minutes.
Population: As only 1 participant was evaluated, results for PK parameters were not reported for the protection of personal data and to avoid re-identification.
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: PK Parameter: AUClast of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: AUClast was defined as the concentration of drug from time zero to the last observable concentration.Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: PK Parameter: CLss/F of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: CLss/F was defined as apparent oral clearance at steady state after administration of the drug. CLss/F = Dose/AUCtau, where "Dose" is the dose of the drug. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: PK Parameter: t1/2 of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: t1/2 was defined as the estimate of the terminal elimination half-life of the drug. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: PK Parameter: Vz/F of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Vz/F was defined as the apparent volume of distribution of the drug. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: PK Parameter: Cmax of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Cmax was defined as the maximum observed concentration of drug.Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: PK Parameter: Tmax of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Tmax was defined as the time (observed time point) of Cmax. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Groups:
- RDV, Part B: Participants received inhaled RDV 62 mg administered as an aerosolized solution by inhalation through facemask daily for 5 days.
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: PK Parameter: Clast of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Clast was defined as the last observable concentration of drug. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: PK Parameter: Tlast of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Tlast was defined as the time (observed time point) of Clast. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: PK Parameter: AUCtau of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: AUCtau is defined as concentration of drug over time (the area under the concentration versus time curve over the dosing interval). Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: PK Parameter: λz of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: λz was defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: PK Parameter: Ctau of RDV and Its Metabolites (GS-441524 and GS-704277) in Parts A and B
Description: Ctau was defined as the observed drug concentration at the end of the dosing interval. Time Frame for PK samples: Sparse PK (all participants): Day 1 (end of nebulization, and optional 2-hour post nebulization), and Day 3 (predose and end of nebulization); Intensive PK (Up to 6 participants/group in Part A & Part B): Day 1 and an additional sample at Day 3 or Day 5 at the following time points: 0 (predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, and 24 hours post end of nebulization.
Time Frame: as for outcome 10
Population: as for outcome 10
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Change in Nasopharyngeal SARS-CoV-2 Viral Load From Baseline to Day 5
Time Frame: Baseline, Day 5
Population: Participants in the Nasopharyngeal mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 11 | 11 | 8 | 9 | 12 | 40 | 12
log10 copies/mL | -2.44 (1.240) | -1.67 (0.992) | -1.78 (1.357) | -1.53 (1.063) | -1.68 (1.475) | -2.09 (1.052) | -2.01 (1.402) | -2.06 (1.321)

23. Secondary Outcome: Change in Oropharyngeal SARS-CoV-2 Viral Load From Baseline to Day 5
Time Frame: Baseline, Day 5
Population: Participants in the Oropharyngeal mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 10 | 11 | 8 | 9 | 9 | 40 | 12
log10 copies/mL | -1.24 (0.957) | -0.88 (0.839) | -1.26 (1.418) | -1.29 (1.457) | -1.13 (1.394) | -1.10 (0.988) | -0.92 (1.213) | -0.66 (1.581)

24. Secondary Outcome: Change in Saliva SARS-CoV-2 Viral Load From Baseline to Day 5
Time Frame: Baseline, Day 5
Population: Participants in the Saliva mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 7 | 10 | 42 | 14
log10 copies/mL | -0.99 (0.562) | -1.26 (1.288) | -0.77 (1.449) | -1.60 (1.443) | -0.31 (0.708) | -0.92 (1.040) | -1.36 (1.056) | -1.15 (0.962)

25. Secondary Outcome: Change in Nasopharyngeal SARS-CoV-2 Viral Load From Baseline to Day 7
Time Frame: Baseline, Day 7
Population: Participants in the Nasopharyngeal mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 9 | 11 | 8 | 10 | 10 | 39 | 15
log10 copies/mL | -3.05 (1.225) | -2.12 (1.051) | -2.09 (1.331) | -1.80 (1.389) | -2.30 (1.257) | -2.34 (1.873) | -2.64 (1.299) | -2.62 (1.555)

26. Secondary Outcome: Change in Oropharyngeal SARS-CoV-2 Viral Load From Baseline to Day 7
Time Frame: Baseline, Day 7
Population: Participants in the Oropharyngeal mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 9 | 10 | 8 | 9 | 9 | 36 | 10
log10copies/mL | -1.76 (1.113) | -0.40 (1.049) | -1.98 (0.971) | -1.73 (1.513) | -1.08 (1.160) | -1.27 (0.845) | -1.07 (1.122) | -0.62 (1.606)

27. Secondary Outcome: Change in Saliva SARS-CoV-2 Viral Load From Baseline to Day 7
Time Frame: Baseline, Day 7
Population: Participants in the Saliva mFAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 10 | 8 | 7 | 8 | 9 | 8 | 38 | 15
log10 copies/mL | -1.28 (1.102) | -1.24 (2.108) | -0.62 (1.406) | -1.91 (1.667) | -0.99 (0.943) | -1.53 (1.553) | -1.69 (1.302) | -1.31 (1.752)

28. Secondary Outcome: Change in Nasopharyngeal SARS-CoV-2 Viral Load From Baseline to Day 14 in Parts A and B
Time Frame: Baseline, Day 14
Population: Participants in the Nasopharyngeal mFAS with available were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 11 | 10 | 8 | 6 | 9 | 11
log10 copies/mL | -4.11 (1.304) | -2.96 (1.475) | -3.31 (1.198) | -2.82 (1.888) | -2.86 (1.837) | -3.41 (1.442)

29. Secondary Outcome: Change in Oropharyngeal SARS-CoV-2 Viral Load From Baseline to Day 14 in Parts A and B
Time Frame: Baseline, Day 14
Population: Participants in the Oropharyngeal mFAS with available were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 10 | 10 | 11 | 6 | 7 | 8
log10 copies/mL | -2.46 (0.908) | -1.47 (0.841) | -2.36 (0.951) | -1.46 (1.194) | -1.95 (1.283) | -2.05 (1.092)

30. Secondary Outcome: Change in Saliva SARS-CoV-2 Viral Load From Baseline to Day 14 in Parts A and B
Time Frame: Baseline, Day 14
Population: Participants in the Saliva mFAS with available were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B
Number analyzed (Participants) | 9 | 8 | 6 | 6 | 8 | 3
log10 copies/mL | -2.58 (1.413) | -2.27 (1.136) | -1.78 (0.618) | -2.30 (1.505) | -2.11 (1.171) | -3.53 (1.253)

31. Secondary Outcome: Time to Negative Nasopharyngeal SARS-CoV-2 Polymerase Chain Reaction (PCR)
Description: The time to negative nasopharyngeal SARS-CoV-2 PCR was defined as the number of days to first confirmed negative (first date of two consecutive dates achieving negative result) using nasopharyngeal sample. Time to negative nasopharyngeal SARS-CoV-2 PCR was calculated using Kaplan-Meier estimates.
Time Frame: Baseline up to Day 17
Population: Participants in the Nasopharyngeal mFAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 11 | 11 | 8 | 10 | 13 | 46 | 16
days | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 17.0 [16.0 to 17.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 16.0 [7.0 to 16.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated.

32. Secondary Outcome: Time to Negative Oropharyngeal SARS-CoV-2 Polymerase Chain Reaction (PCR)
Description: The time to negative oropharyngeal SARS-CoV-2 PCR was defined as the number of days to first confirmed negative (first date of two consecutive dates achieving negative result) using an oropharyngeal sample. Time to negative oropharyngeal SARS-CoV-2 PCR was calculated using Kaplan-Meier estimates.
Time Frame: Baseline up to Day 17
Population: Participants in the Oropharyngeal mFAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 11 | 41 | 12
days | 14.0 [5.0 to 15.0] | 15.0 [4.0 to 16.0] | 13.0 [7.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated. | 5.0 [2.0 to 15.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 14.0 [5.0 to 15.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated.

33. Secondary Outcome: Time to Negative Saliva SARS-CoV-2 Polymerase Chain Reaction (PCR)
Description: The time to saliva SARS-CoV-2 PCR was defined as the number of days to first confirmed negative (first date of two consecutive dates achieving negative result) using saliva sample. Time to negative saliva SARS-CoV-2 PCR was calculated using Kaplan-Meier estimates.
Time Frame: Baseline up to Day 17
Population: Participants in the Saliva mFAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 11 | 10 | 8 | 10 | 9 | 12 | 45 | 16
days | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 17.0 [13.0 to 17.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 16.0 [7.0 to 16.0] | 14.0 [3.0 to 15.0] | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants had negative SARS-CoV-2 PCR result, the median time to negative SARS-CoV-2 PCR couldn't be calculated. | 16.0 [7.0 to 16.0]

34. Secondary Outcome: Time to Alleviation (Mild or Absent) of Baseline COVID-19 Symptoms as Reported on the COVID-19 Adapted InFLUenza Patient-Reported Outcome (FLU-PRO©) Questionnaire in Part C
Description: The InFLUenza Patient-Reported Outcome (FLU-PRO©) is a 32-item patient-reported outcome questionnaire that assesses the severity of symptoms of influenza and influenza-like illness across six body systems. An additional two items can be added to assess changes in taste or smell, if the instrument is used to quantify symptoms in studies of COVID-19. Each domain scores ranges from 0 (symptom-free) to 4 (very severe symptoms). Higher scores on this scale represent higher disease severity. Alleviation is defined as symptom scores as 2 or higher at baseline are scored as 0 (absent) or 1 (mild) at post-baseline, and symptoms scored as 1 at baseline are scored as 0 at post-baseline, and for two consecutive days. Time to alleviation was calculated using Kaplan-Meier estimates.
Time Frame: First dose date up to Day 14
Population: Participants in FAS with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RDV, Part C | Placebo, Part C
Number analyzed (Participants) | 39 | 9
days | NA [NA to NA] — Since less than 50% of participants achieved alleviation, the median time to alleviation couldn't be calculated. | NA [NA to NA] — Since less than 50% of participants achieved alleviation, the median time to alleviation couldn't be calculated.

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 5 days plus 30 days All-Cause Mortality: Randomization date up to 35 days
Description: Adverse Events: The Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study treatment.
  All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Arm/Group | RDV, Part A | RDV + Placebo, Part A | Placebo, Part A | RDV, Part B | RDV + Placebo, Part B | Placebo, Part B | RDV, Part C | Placebo, Part C
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/12 | 0/12 | 0/12 | 0/13 | 0/62 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 2/12 | 0/12 | 1/12 | 1/13 | 0/61 | 0/20
Other Adverse Events (participants affected / at risk) | 7/12 | 7/12 | 5/12 | 4/12 | 6/12 | 5/13 | 24/61 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RDV, Part A (N=12) | RDV + Placebo, Part A (N=12) | Placebo, Part A (N=12) | RDV, Part B (N=12) | RDV + Placebo, Part B (N=12) | Placebo, Part B (N=13) | RDV, Part C (N=61) | Placebo, Part C (N=20)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RDV, Part A (N=12) | RDV + Placebo, Part A (N=12) | Placebo, Part A (N=12) | RDV, Part B (N=12) | RDV + Placebo, Part B (N=12) | Placebo, Part B (N=13) | RDV, Part C (N=61) | Placebo, Part C (N=20)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT04539262/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT04539262/SAP_001.pdf